CLINICAL TRIAL: NCT06534281
Title: Pilot Study of Multi-Branch AOrtic Reconstruction With G-iliac System (BAO-G) Technique in Thoracoabdominal Aortic Aneurysm Endovascular Repair
Brief Title: Pilot Study of BAO-G Technique in TAAA Endovascular Repair
Status: Enrolling by invitation | Phase: Early Phase 1 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Liu Bao, Professor, Peking Union Medical College Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BAO-G-01
Record Dates: First submitted 2024-07-29; First posted 2024-08-02 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-08

CONDITIONS: Aortic Aneurysm, Thoracoabdominal
Keywords: BAO-G technique; thoracoabdominal aortic aneurysm; iliac-branched devices; endovascular repair
MeSH Terms: conditions — Aortic Aneurysm, Thoracoabdominal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BAO-G group (Experimental)
  Interventions: Procedure: BAO-G

INTERVENTIONS:
Procedure: BAO-G — Using G-iliac system to reconstruct the visceral branches of in endovascular repair of thoracoabdominal aortic aneurysm.

SUMMARY:
Multi-Branch AOrtic Reconstruction With G-iliac System (BAO-G) Technique is a novel technique of endovascular repair of thoracoabdominal aortic aneurysm, which using off-the-shelf iliac branched devices to reconstruct the visceral branches. This study aims to evaluate the safety and efficacy of BAO-G in thoracoabdominal aortic aneurysm endovascular repair.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with TAAA, confirmed by aortic CTA.
2. TAAA diameter ≥ 6cm, or symptomatic TAAA with diameter ≥ 4cm.
3. Informed consent signed.

Exclusion Criteria:

1. were pregnant.
2. had a history of previous endovascular or open repair.
3. had other contraindications of endovascular treatment.
4. Uncontrolled autoimmune disease.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2035-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of visceral branch patency | Month 0, 3, 6, 12, and annually after surgery
  the patency of visceral branches measured by radiological test
Incidence of endoleak | Month 0, 3, 6, 12, and annually after surgery
  The incidence of endoleak measured by radiological test
Incidence of re-operation | Month 0, 3, 6, 12, and annually after surgery
  The incidence of re-operation for any adverse events, confirmed by medical record and outpatient follow up

SECONDARY OUTCOMES:
Incidence of organ ischemia | Month 0, 3, 6, 12, and annually after surgery
  Incidence of organ ischemia, measured by physical examination and radiological test
Incidence of acute kidney injury | perioperative period
  The incidence of acute kidney injury, measured by serum creatinine level
Incidence of acute liver function injury | perioperative period
  The incidence of acute liver function injury, measured by serum transaminase level
Incidence of acute pancreatitis | perioperative period
  The incidence of acute pancreatitis, measured by serum amylase level

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No